CLINICAL TRIAL: NCT02495259
Title: Comparison of Placement of Double-lumen Endobronchial Tube Using GlideScope With 2 Different Stylet Configurations vs Standard Macintosh Laryngoscopy
Brief Title: Comparison of Double Lumen Tube Placement Techniques
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI is leaving the institution
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Igor Zhukov, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB00081067
Record Dates: First submitted 2015-07-09; First posted 2015-07-13 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-07-27 (Actual); Status verified 2018-06

CONDITIONS: Airway Morbidity; Intubation Complication; Tracheal Intubation Morbidity; Anesthesia Intubation Complication; Failed or Difficult Intubation, Sequela
Keywords: Double-lumen endobronchial tube; Laryngoscopy; intubating stylet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ZU-bend stylet with GlideScope technique (Experimental): Subjects scheduled for thoracic surgery in which the surgeon requests lung isolation will undergo laryngoscopy and intubation using the ZU-bend with the GlideScope technique of a double lumen endobronchial tube (DLT) placement as part of the anesthesia procedure prior to surgery.
  Interventions: Device: ZU-bend stylet; Device: GlideScope
- GlideScope with the GlideRite stylet (Active Comparator): Subjects scheduled for thoracic surgery in which the surgeon requests lung isolation will undergo laryngoscopy and intubation using the GlideScope with the GlideRite stylet for placement of a double lumen endobronchial tube (DLT) as part of the anesthesia procedure prior to surgery.
  Interventions: Device: GlideScope; Device: GlideRite stylet
- Macintosh blade and a regular DLT stylet (Active Comparator): Subjects scheduled for thoracic surgery in which the surgeon requests lung isolation will undergo laryngoscopy and intubation using the direct laryngoscopy technique with the Macintosh blade and a regular double lumen endobronchial tube (DLT) stylet as part of the anesthesia procedure prior to surgery.
  Interventions: Device: Macintosh blade; Device: Regular Double-lumen endobronchial tube (DLT) Stylet

INTERVENTIONS:
Device: ZU-bend stylet — Laryngoscopy and intubation after induction of anesthesia will be done using the GlideScope and the ZU-bend stylet. The ZU-bend is a specific shaping technique of the intubating stylet that is closely related to the GlideScope blade curvature. Zu-bend stylet is withdrawn as a part of placement procedure during the DLT advancement. Thereafter, GlideScope is removed and placement of the double-lumen endobronchial tube is verified with capnography and fiberoptic bronchoscopy in the usual manner.
  Arms: ZU-bend stylet with GlideScope technique
Device: GlideScope — Laryngoscopy and intubation after induction of anesthesia will be done using the the GlideScope technique. The GlideScope is a video laryngoscope that provides a real-time view of the airway and tube placement during intubation. GlideScope is removed after DLT is in the trachea, and placement of the double-lumen endobronchial tube is verified with capnography and fiberoptic bronchoscopy in the usual manner.
  Arms: GlideScope with the GlideRite stylet; ZU-bend stylet with GlideScope technique
Device: GlideRite stylet — Laryngoscopy and intubation after induction of anesthesia will be done with the GlideScope using the GlideRite stylet. The GlideRite stylet is specifically designed to work with the GlideScope and provides the necessary rigidity and curvature to an otherwise flexible tube. GlideRite stylet is withdrawn as a part of placement procedure during the DLT advancement. Thereafter, GlideScope is removed and placement of the double-lumen endobronchial tube is verified with capnography and fiberoptic bronchoscopy in the usual manner.
  Arms: GlideScope with the GlideRite stylet
Device: Macintosh blade — Direct laryngoscopy and intubation after induction of anesthesia will be done with the Macintosh blade and a regular double-lumen endobronchial tube (DLT) stylet. The Macintosh blade is used to facilitate visualization of the larynx during double or single lumen endobronchial tube placement. After intubation the Macintosh laryngoscope is removed and the confirmation of the successful placement of the double-lumen endobronchial tube in done in the standard fashion.
  Other Names: Laryngoscope blade
  Arms: Macintosh blade and a regular DLT stylet
Device: Regular Double-lumen endobronchial tube (DLT) Stylet — Direct laryngoscopy and intubation after induction of anesthesia will be done with a regular double-lumen endobronchial tube (DLT) stylet and the Macintosh blade. The DLT stylet is withdrawn as a part of placement procedure during the DLT advancement. Thereafter, Macintosh laryngoscope is removed and placement of the double-lumen endobronchial tube is verified with capnography and fiberoptic bronchoscopy in the usual manner.
  Arms: Macintosh blade and a regular DLT stylet

SUMMARY:
The purpose of this study is to compare three different standard of care methods of double-lumen endobronchial tube (DLT) placement in patients who are scheduled to have thoracic surgery in which lung isolation is required.

DETAILED DESCRIPTION:
The purpose of this study is to compare three different standard of care methods of double-lumen endobronchial tube (DLT) placement in patients who are scheduled to have thoracic surgery in which lung isolation is required. The investigators want to evaluate the technique of placement of the double-lumen endobronchial tube (DLT) using an included stylet that has been radically bent (ZU-bend) as compared to a commercial GlideRite stylet with the GlideScope and direct laryngoscopy using the Macintosh laryngoscope. A double-lumen endobronchial tube (DLT) is a breathing tube utilized to manage the airway when lung separation is needed for a surgical procedure. The investigator wants to evaluate how long it takes for successful placement of the double-lumen endobronchial tube (DLT) and assess the difficulty of the procedure experienced by the physician performing the intubation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients requiring a double-lumen endobronchial tube placement for surgery at Emory University Hospital or Emory University Hospital Midtown
2. Patients willing and able to provide written informed consent

Exclusion Criteria:

1. Patients in whom a previously difficult airway manipulation was recorded on an anesthetic record
2. Lung transplantation procedures, as underlying pulmonary disorder that will confound the SpO2 (peripheral capillary oxygen saturation) metric
3. Any patient who is receiving anticoagulants in excess of a daily aspirin, patients with an International Normalized Ratio or INR >1
4. Patients in whom one lung ventilation or placement of a double-lumen endobronchial tube is contraindicated
5. Patients who require a rapid-sequence intubation
6. Patients undergoing emergency procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07-27 (Actual); Study Completion 2017-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Zhukov, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
Started | 7 | 4 | 8
Completed | 7 | 3 | 8
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet | Total
Number analyzed (Participants) | 7 | 4 | 8 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 4 | 10
  >=65 years | 4 | 1 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 6 | 11
  Male | 4 | 2 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 6 | 2 | 6 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 4 | 8 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Time to Place the Double-lumen Endobronchial Tube
Description: The time taken for successful intubation will be recorded by the anesthetist. The total duration from the time the laryngoscope is placed at the patient's lips to the first detection of End-tidal CO2 (EtCO2), an average of 120 seconds, will be recorded in seconds. A higher duration noted is indicative of a longer time taken for successful intubation. 0 seconds (laryngoscope at patient's lips), (first End-tidal CO2 (EtCO2) detection)
Time Frame: during laryngoscope placement, up to 120 seconds
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
Number analyzed (Participants) | 7 | 3 | 8
sec | 111 (44.9) | 54 (13.1) | 55 (17.5)

2. Secondary Outcome: Success Rate of First Endobronchial Intubation Attempt
Description: The rate of first intubation attempt success will be recorded by the anesthetist. A successful first attempt intubation is when the double-lumen endobronchial tube is placed during the initial laryngoscopy within 120 seconds. The average time for successful intubation is 120 seconds, which is the time from when the laryngoscope is placed at the patient's lips to the first detection of End-tidal CO2 (EtCO2). Higher numbers of successful first attempt intubations indicate better rates of success of first endobronchial intubation attempts .
Time Frame: during laryngoscope placement, up to 120 seconds
Measure: Count of Participants; unit: Participants
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
Number analyzed (Participants) | 7 | 3 | 8
Participants | 4 | 3 | 8

3. Secondary Outcome: Assessment of Difficulty of Intubation
Description: The ease of successful placement of the double-lumen endobronchial tube (DLT) will be assessed by the anesthetist's responses to a multi-question form which includes the following items that are scored; overall ease of intubation, laryngoscope insertion, glottic view, double-lumen endobronchial tube (DLT) delivery and placement. The subjective scores range from 0-10; where 0=worst, 10=best. The average time for successful intubation is 120 seconds, which is the time from when the laryngoscope is placed at the patient's lips to the first detection of End-tidal CO2 (EtCO2).
Time Frame: during laryngoscope placement, up to 120 seconds
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
Number analyzed (Participants) | 7 | 3 | 8
units on a scale | 8 (1.8) | 10 (0) | 2 (2.2)

4. Secondary Outcome: Number of Cases With Complications
Description: Number of cases with complications during intubation will be will be assessed by the anesthetist's responses to a multi-question form which includes the following items; blood on device, SpO2 (peripheral capillary oxygen saturation) <96%, lip and dental trauma and double-lumen endobronchial tube (DLT) cuff rupture. The responses are recorded as Yes or No for each item. A 'yes' response indicates a complication. The average time for successful intubation is 120 seconds, which is the time from when the laryngoscope is placed at the patient's lips to the first detection of End-tidal CO2 (EtCO2).
Time Frame: during laryngoscope placement, up to 120 seconds
Measure: Number; unit: cases of complications
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
Number analyzed (Participants) | 7 | 3 | 8
cases of complications | 0 | 0 | 0

5. Secondary Outcome: Number of Cases of Voice Change
Description: Any voice change in the patient after extubation will be assessed in the Post-Operative Admission Unit (PACU) by asking the patient if any change in voice is experienced (Yes/No). The subjective answer given by the patient will be recorded. The average time for the patient to sufficiently recover to respond is expected to be 60 minutes after extubation.
Time Frame: Up to 60 minutes after extubation
Measure: Number; unit: cases of voice change
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
Number analyzed (Participants) | 7 | 3 | 8
cases of voice change | 3 | 1 | 2

6. Secondary Outcome: Throat Pain
Description: Any voice change in the patient after extubation will be assessed in the Post-Operative Admission Unit (PACU) by recording the patient's response to the degree of pain experienced. An analog pain scale will be used for scoring where: 0= no pain and 10= severe pain. The average time for the patient to sufficiently recover to respond is expected to be 60 minutes after extubation.
Time Frame: Up to 60 minutes after extubation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
Number analyzed (Participants) | 7 | 3 | 8
units on a scale | 1.4 (1.6) | 1.3 (1.5) | 1.9 (2.2)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | ZU-bend Stylet With GlideScope Technique | GlideScope With the GlideRite Stylet | Macintosh Blade and a Regular DLT Stylet
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/4 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/4 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT02495259/Prot_SAP_000.pdf